CLINICAL TRIAL: NCT00004238
Title: A Phase II Study of 10-Propargyl-10-Deazaaminopterin (PDX) in Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: 10-Propargyl-10-Deazaaminopterin in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-053; CDR0000067482 (Registry Identifier: PDQ (Physician Data Query)); NCI-H99-0045
Record Dates: First submitted 2000-01-28; First posted 2004-04-12 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — 10-propargyl-10-deazaaminopterin

INTERVENTIONS:
Drug: pralatrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of 10-propargyl-10-deazaaminopterin in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine objective response rate, duration of response, and time to disease progression in patients with stage IIIB (pleural or pericardial disease) or stage IV non-small cell lung cancer treated with 10-propargyl-10-deazaaminopterin as first line or second line chemotherapy. II. Determine the toxicity of this drug in this patient population. III. Determine duration of survival in these patients. IV. Determine quality of life of these patients.

OUTLINE: Patients receive 10-propargyl-10-deazaaminopterin IV on days 1 and 15. Treatment repeats every 4 weeks in the absence of unacceptable toxicity or disease progression. Quality of life is assessed at the beginning of each course. Patients are followed every 8 weeks for disease progression.

PROJECTED ACCRUAL: A total of 19-39 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage IIIB (pleural or pericardial disease) or stage IV non-small cell lung cancer Measurable or evaluable indicator lesion that has not been irradiated Pleural effusions, bone metastases, brain metastases, elevated serum enzymes, and abnormal radionucliotide scans are unacceptable as sole indicator lesions No clinically significant pleural effusions or ascites No grade III or IV edema No prior pneumonectomy No symptomatic or uncontrolled brain or leptomeningeal involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: WBC at least 4,000/mm3 Hemoglobin at least 10 g/dL Platelet count at least 160,000/mm3 Hepatic: Bilirubin no greater than 1.0 mg/dL AST no greater than 1.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 5 times ULN Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 50 mL/min Cardiovascular: No unstable cardiac disease requiring treatment Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No other concurrent active cancer No history of significant neurologic or psychiatric disorders, including psychotic disorders, dementia, or seizures No active uncontrolled infection No other serious illness or medical condition

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy OR Progression after stable disease or initial response to 1 prior chemotherapy regimen, including 1 preoperative or adjuvant chemotherapy regimen Endocrine therapy: Concurrent steroids allowed if dose is stable Radiotherapy: See Disease Characteristics At least 3 weeks since prior radiotherapy Surgery: See Disease Characteristics Other: No prior antifolates At least 7 days since prior folic acid supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Krug, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Krug LM, Azzoli CG, Kris MG, Miller VA, Khokhar NZ, Tong W, Ginsberg MS, Venkatraman E, Tyson L, Pizzo B, Baez V, Ng KK, Sirotnak FM. 10-propargyl-10-deazaaminopterin: an antifolate with activity in patients with previously treated non-small cell lung cancer. Clin Cancer Res. 2003 Jun;9(6):2072-8. PMID 12796370